CLINICAL TRIAL: NCT05164042
Title: Allogeneic CD19 CAR-T Cells for the Treatment of Relapsed/Refractory B-cell Acute Lymphoblastic Leukemia
Acronym: CAR-T
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen University General Hospital (Other)
Responsible Party: Principal Investigator, YuLi, Professor, Shenzhen University General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEM-ONCO-007
Record Dates: First submitted 2021-11-22; First posted 2021-12-20 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-02

CONDITIONS: Relapse Leukemia; Refractory Leukemia
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Subjects who meet the enrollment conditions will receive intravenous infusion of allogeneic CD19 CAR-T cells after pretreatment.
  Interventions: Biological: Allogeneic CD19 CAR-T cells

INTERVENTIONS:
Biological: Allogeneic CD19 CAR-T cells — infusion of allogeneic CD19 CAR-T cells

SUMMARY:
CD19 CAR-T has been widely developed in patients with R/R ALL and has also been generally recognized by the industry. In 2017, the U.S. FDA approved Novartis's CD 19 CAR-T product Kymriah for the treatment of R/R ALL. However, these CAR-T cells are constructed from patients' autologous T cells, and the production and preparation time is long; on the other hand, most patients have received multiple chemotherapy before CAR-T treatment, and the quantity and quality of T cells often cannot meet the needs of clinical treatment. It is also an important factor leading to the failure of CAR-T cell therapy, which limits the large-scale clinical application of CAR-T.

T cells derived from healthy donors are not only sufficient in quantity and quality guaranteed, but also available at any time. In December 2020, lancet reported a clinical study of 19 patients receiving allogeneic CAR-T cell ALL. 14 patients were evaluated as CR/CRi (67%) 28 days after treatment, and the median sustained remission time was 4.1 moon. Allogeneic CAR-T cells are safe and effective for the treatment of ALL, and their clinical application range is expected to improve the remission rate and survival rate of patients with R/R ALL.

DETAILED DESCRIPTION:
Chimeric antigen receptor (CAR) T cells enable T cells to recognize and kill tumor cells that express specific antigens through genetic engineering. CD19 is expressed on the membrane surface of pre-B cells and mature B cells, but not on the surface of T cells and normal granulocytes. It is an ideal therapeutic target for B cell-derived tumors. A large number of previous studies have confirmed that CD19 CAR-T cells are a safe and effective method for the treatment of ALL. In 2018, New England Journal published the long-term follow-up data of CD19 CAR-T for relapse/refractory (R/R) ALL, 53 patients with r/r ALL who received a single infusion of CD19 CAR-T The response efficiency (CR+PR) reached 98%, of which about 83% of CR patients, with a median survival time of 12.9 months; greatly improved the remission rate and survival rate of r/r ALL patients.

Nowadays,CD19 CAR-T has been widely developed in patients with R/R ALL and has also been generally recognized by the industry. In 2017, the U.S. FDA approved Novartis's CD CAR-T product Kymriah for the treatment of R/R ALL. However, these CAR-T cells are constructed from patients' autologous T cells, and the production and preparation time is long; on the other hand, most patients have received multiple chemotherapy before CAR-T treatment, and the quantity and quality of T cells often cannot meet the needs of clinical treatment. It is also an important factor leading to the failure of CAR-T cell therapy, which limits the large-scale clinical application of CAR-T.

T cells derived from healthy donors are not only sufficient in quantity and quality guaranteed, but also available at any time. In December 2020, lancet reported a clinical study of 19 patients receiving allogeneic CAR-T cell ALL. 14 patients were evaluated as CR/CRi (67%) 28 days after treatment, and the median sustained remission time was 4.1 moon. Allogeneic CAR-T cells are safe and effective for the treatment of ALL, and their clinical application range is expected to improve the remission rate and survival rate of patients with R/R ALL.

ELIGIBILITY:
Inclusion Criteria:

1. 14-70 years old (including 14, 70 years old), no gender limit;
2. According to the 2020 World Health Organization (WHO) diagnostic criteria, it is diagnosed as relapsed/refractory B-cell acute lymphoblastic leukemia (r/r B-ALL);
3. The ECOG behavior status score is 0-2 points;
4. Expected survival time ≥ 3 months;
5. Flow cytometry confirms that the original cells express CD19;
6. Those who have failed autologous CAR-T cell preparation or autologous CAR-T cell therapy under the existing technical conditions;
7. No serious heart, lung, liver, or kidney disease;
8. Ability to understand and willing to sign the informed consent form for this trial.

Exclusion Criteria:

1. Primitive cells do not express CD19;
2. Active infection;
3. Abnormal liver function (total bilirubin>1.5×ULN, ALT>2.5×ULN), abnormal renal function (serum creatinine>1.5×ULN);
4. People with unstable angina or New York Heart Association class 3/4 congestive heart failure, multiple organ dysfunction;
5. HIV/AIDS patients;
6. Those who need long-term anticoagulation (warfarin or heparin), antiplatelet (aspirin, dose>300mg/d; clopidogrel, dose>75mg/d) treatment;
7. Those who received radiotherapy within 4 weeks before the start of the study;
8. Known or suspected drug abuse or alcohol dependence;
9. People with mental illness or other conditions cannot obtain informed consent, and cannot cooperate with the requirements of completing the experimental treatment and inspection procedures;
10. Participated in other clinical trials within 30 days;
11. Pregnant or lactating women, male subjects (or their partners) or female subjects have a pregnancy plan during the study period to 6 months after the end of the test, and are unwilling to use a medically approved effective contraceptive measure during the test period (Such as intrauterine contraceptive devices or condoms);
12. Those who are judged by the investigator to be unsuitable to participate in this trial.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
CRR | From data of enrollment until the first documented progression of disease, up to 2 years.
  Complete remission rate

SECONDARY OUTCOMES:
OS | From admission to the end of follow up, up to 2 years.
  Overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Li Yu, Dr, Principal Investigator — Shenzhen University General Hospital
Locations (1):
- Li Yu, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No